CLINICAL TRIAL: NCT02498275
Title: Effect of RO6871765 and RO7011785 on Immune Response With the Stimulation of Peripheral Blood Mononuclear Cells (PBMCs) in Chinese Healthy Volunteers and Chronic Hepatitis B Patients
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: YP29018
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Healthy volunteers: Blood samples from healthy volunteers will be collected for ex vivo stimulation and for further sample preparation and analysis.
- Nucleoside/nucleotide analogue-treated CHB patients: Blood samples from nucleoside/nucleotide analogue-treated CHB patients will be collected for ex vivo stimulation and for further sample preparation and analysis.
- Treatment-naive CHB patients: Blood samples from treatment-naïve CHB patients will be collected for ex vivo stimulation and for further sample preparation and analysis.

SUMMARY:
This is an exploratory study to characterize the ex vivo immune response to RO6871765 or RO7011785 stimulation of peripheral blood mononuclear cells (PBMCs) extracted from healthy volunteers and chronic hepatitis B (CHB) patients.

ELIGIBILITY:
Inclusion Criteria:

All population:

* Chinese population
* Adequate hematological function: platelet count greater than or equal to (>=) 100*10^9 per liter (/L), hemoglobin (Hb) >= 12 grams/deciliter (g/dL) (male) or >= 11 g/dL (female), white blood cell (WBC) count >= 4*10^9/L and <= 11*10^9/L

Healthy volunteers:

* Absence of evidence of any active or chronic disease
* Negative hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb), hepatitis B envelope antigen (HBeAg), hepatitis B envelope antiody (HBeAb) and hepatitis B core antibody (HBcAb)
* Adequate liver function: transaminases alanine aminotransferase (ALT) <= 1.0 times the upper limit of normal (ULN)

Treatment naïve CHB patients:

* HBsAg-positive (>=250 international unit/milliliter [IU/mL]), compensated liver function, non-cirrhotic
* HBeAg-positive, HBV DNA >= 200,000 IU/ml or equivalent copies/mL, ALT >1.5 times the ULN and ALT <8 times the ULN

HBeAg-negative nucleoside/nucleotide analogue-treated CHB patients:

* Subjects who HBeAg-seroconverted on nucleoside/nucleotide analogue therapy (treatment for 1 to 3 years prior to enrollment) with HBV DNA <90 IU/mL or below a detection level acceptable by both the sponsor and investigator for at least the preceding 6 months; HBeAg negative and HBeAb positive
* HBsAg-positive (>=250 IU/mL), compensated liver function, non-cirrhotic -ALT <= 1*ULN

Exclusion Criteria:

* Use of steroids or other immune suppressive agents within the last 4 weeks that would impact the number/functions of white blood cells (WBC)
* Any other diseases or clinical laboratory finding giving reasonable suspicion of a disease or condition (including, but not limited to, cancer, lupus erythematosus, rheumatoid arthritis, or other autoimmune disease) that could confound the result of the study
* Positive Hepatitis A immunoglobulin M (IgM) antibody, Hepatitis C antibody (HCV Ab) or human immunodeficiency virus (HIV) at screening
* Significant acute infection, example; influenza, acute gastrointestinal symptoms or any other clinically significant illness within 2 weeks
* Previous/concurrent treatment with interferon-based therapy for CHB

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese population: healthy volunteers, treatment naive CHB patients and nucleoside or nucleotide analogue treated CHB patients
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Correlation coefficients between baseline toll-like receptor 7 (TLR7) expression and ex vivo immune response upon stimulation of PBMCs with RO6871765 or RO7011785 (in terms of cytokine release and gene expression) | Day 1
Cytokine/chemokine production | Day 1
Induction of interferon-responsive genes | Day 1

SECONDARY OUTCOMES:
Number or percentages of T-lymphocytes in healthy volunteers and subjects with CHB | Screening Up to Day 1
Number or percentages of B-lymphocytes in healthy volunteers and subjects with CHB | Screening up to Day 1
Number or percentages of natural killer (NK) -cells in healthy volunteers and subjects with CHB | Screening up to Day 1
Number or percentages of myeloid dendritic cells (mDCs) in healthy volunteers and subjects with CHB | Screening up to Day 1
Number or percentages of plasmacytoid dendritic cells (pDCs) in healthy volunteers and subjects with CHB | Screening up to Day 1
Ex-vivo antiviral activity of PBMC supernatant | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Shanghai, China